CLINICAL TRIAL: NCT03248856
Title: Triamcinolone Levels in Cochlear Perilymph
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christoph Arnoldner (Other)
Responsible Party: Sponsor-Investigator, Christoph Arnoldner, Assoc Prof PD Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1456/2017; 2017-002377-19 (EudraCT Number)
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Other): Group 1 will receive triamcinolone acetonide 10mg 20 to 24hours before sampling.
  Interventions: Drug: Triamcinolone Acetonide
- Group 2 (Other): Group 2 will receive triamcinolone acetonide 40mg 20 to 24hours before sampling.
  Interventions: Drug: Triamcinolone Acetonide
- Group 3 (Other): Group 3 will receive triamcinolone acetonide 10mg 1 to 2 hours before sampling.
  Interventions: Drug: Triamcinolone Acetonide
- Group 4 (Other): Group 3 will receive triamcinolone acetonide 40mg 1 to 2 hours before sampling.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Intratympanic administration

SUMMARY:
In this study Triamcinolone acetonide will be applied intratympanically before cochlear implant surgery. After round window exposure, a perilymph sample and simultaneously a blood sample will be drawn. Triamcinolone levels will then be analyzed in the samples.

DETAILED DESCRIPTION:
At the ENT department of the university hospital Vienna (AKH Wien) patients are treated with intratympanic triamcinolone acetonide before cochlea implantation to reduce inflammation and in some cases to protect residual hearing. Triamcinolone acetonide levels in cochlear perilymph will be evaluated in an open prospective clinical study. Patients scheduled for cochlear implant surgery between 18 and 90 years will be included. Patients who are treated with steroids preoperatively will be excluded from the study. Patients will be randomized after inclusion to one of four groups. The randomization is carried out to generate hypothesis for the needed dose and best time of application in the future. Triamcinolone acetonide will then be applied 20-24h before surgery or at the beginning of the surgery, depending on randomization (see below). About 20 µl of perilymph will be sampled simultaneously to a blood sample during cochlear implant surgery.

The probes will be stored at -80°C. Triamcinolone acetonide levels of the blood and perilymph will be determined by the pharmaceutical laboratory (Department of Pharmaceutical Technology and Biopharmaceutics, University of Vienna).

The patients will be randomized to 4 groups. Group 1 - Volon A 10mg administration 20 - 24 hours before sampling. Group 2 - Volon A 40mg administration 20 - 24 hours before sampling. Group 3 Volon A 10mg - administration 1 to 2 hours before sampling. Group 4 - Volon A 40mg administration 1 to 2 hours before sampling.

The time interval of application (1 to 2 hours and 20 to 24 hours before sampling) are a result of varying time of surgery depending on surgeons and patient anatomy as well as day to day clinical organization. Patients can withdraw consent at any time of the study.

The active phase of each patient will be between 6 and 9 days depending on time of follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 90 years will be included in the study, who will undergo a cochlear implantation and are willing to participate in the study

Exclusion Criteria:

* Patients younger than 18 years
* Patients who receive cortisone on a regular basis or receive cortisone i.v. or p.o. preoperatively
* Patients with contraindications against the administration of Volon A

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Triamcinolone levels in comparison | 2 years
  Absorption of Triamcinolone acetonide in cochlear perilymph in comparison to dissemination to the blood circulation

SECONDARY OUTCOMES:
Triamcinolone stability | 2 years
  The stability of triamcinolone acetonide levels in the cochlear perilymph
Triamcinolone concentrations | 2 years
  Perilymph concentrations and blood concentrations of triamcinolone acetonide after administration of different Triamcinolone acetonide doses.
Impedances | 2 years
  Difference of impedances of patients receiving different doses at different timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna (AKH), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: January 2020

REFERENCES:
- [Derived] Dahm V, Gausterer JC, Auinger AB, Honeder C, Gabor F, Reznicek G, Kaider A, Riss D, Arnoldner C. Evaluation of Levels of Triamcinolone Acetonide in Human Perilymph and Plasma After Intratympanic Application in Patients Receiving Cochlear Implants: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Nov 1;147(11):974-980. doi: 10.1001/jamaoto.2021.2492. PMID 34591079